CLINICAL TRIAL: NCT01610973
Title: Comparison of Manual and Automated Techniques in Achieving Posterior Lamellar Transplantation of the Cornea
Brief Title: Comparison of Two Techniques in Achieving Corneal Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/084/HP; 2011-A00221-40
Record Dates: First submitted 2012-04-25; First posted 2012-06-04 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Fuch's Endothelial Dystrophy
Keywords: Fuch's dystrophy; Corneal graft
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual preparation (Experimental): Manual preparation of the graft
  Interventions: Procedure: Endothelial descemet membrane graft
- Automatized preparation (Active Comparator): Automatized preparation of the graft with microkeratoma
  Interventions: Procedure: Endothelial descemet membrane graft

INTERVENTIONS:
Procedure: Endothelial descemet membrane graft — Standard Endothelial descemet membrane graft
  Arms: Manual preparation
Procedure: Endothelial descemet membrane graft — Standard Endothelial descemet membrane graft
  Arms: Automatized preparation

SUMMARY:
The cornea is a transparent membrane, half a millimeter thick, embedded as a window in front of the eye.

When the eye becomes opaque, the eye is not seeing and the only way to restore the visual acuity is to replace the cornea by performing a graft (4000 surgeries per year in France). In half the cases the opacification of the cornea is secondary to dysfunction of the endothelium, cell layer of 15 μm thickness, covering its posterior surface, in charge of regulating the moisture of the corneal thickness and therefore its transparency.

While the total corneal transplantation has long been the only intervention for these diseases, it is now possible, from 4-5 years, to replace only the very thin: it is called endothelial transplant or graft lamellar later. This intervention is now experiencing significant success as it reduces very significantly the incidence of complications found after transplantation of total cornea and the visual recovery period. This type of transplant is still difficult to achieve and the best technique is not yet established.

Indeed, posterior lamellar transplantation of the cornea may be done manually or using an automated device. Manual techniques allow the preparation of grafts extremely thin but are difficult to achieve while the automatic techniques, easier, prepare thicker grafts that may be less efficient in visual recovery.

The aim of this project is to conduct a prospective study in order to compare these two techniques in terms of postoperative visual recovery and the vitality of the graft during the first year. To date, there is no such study.

The department of Ophthalmology in the University Hospital of Rouen is one of the most famous French teams in the field of cornea transplants and receives many patients from different French regions. The recruitment of 40 patients needed to study should be done without great difficulty over a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* men and woman
* 18 years old or more
* Patient having been informed about the study and having signed a non-opposition to the participation

Exclusion Criteria:

* Patient presenting an associated eye pathology previously known and able to limit the visual recovery (age-related macular degeneration, diabetic retinopathy, ...)
* Pregnant women, parturient or breast feeding
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Measurement of visual acuity | 1 year

SECONDARY OUTCOMES:
Occular hypertension | Day 7, Day 15, Month 1, Month 2, Month 6, 1 year
  Measurement of occular hypertension
Measurement of visual acuity | Month 1, Month 2, Month 6
Partial or complete graft detachment | Day 7, Day 15, Month 1, Month 2, Month 6, 1 year
  % of detachment
Necessity of air injection | Day 7, Day 15, Month 1, Month 2, Month 6, 1 year
  Necessity of air injection : yes/no
Defeat of the graft | Day 7, Day 15, Month 1, Month 2, Month 6, 1 year
  Defeat of the graft : yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Marc MURAINE, Pr, Principal Investigator — UH Rouen
Locations (1):
- UH Rouen, Rouen, France